CLINICAL TRIAL: NCT04864613
Title: The Importance of ENDING-S Score in the Diagnosis of Palliative Patients in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Cihangir Dogu, Specialist MD, Ankara City Hospital Bilkent
Other Study IDs: 2636
Record Dates: First submitted 2021-01-30; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Palliative Care; Critical Care; Length of Stay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In our study, we aim to predict palliative care patients earlier, to reduce hospitalization periods and to prevent intensive care unit occupation by palliative care patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years will be included in the study. Patients staying longer than 48 hours intensive care will be included in the study.

Exclusion Criteria:

* Patients younger than 18 years. Patients staying less than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Recognition of palliative care unit patients before intensive care discharge | Fourth day of intensive care follow up
  ENDING-S Scoring system used to predict patients who were followed up in intensive care units and discharged to palliative care unit during their hospitalization. We aim to identify patients who are likely to be admitted to palliative care centers following their admission to intensive care units, and to prepare a palliative care center before the discharge from the intensive care.

CONTACTS AND LOCATIONS:
Overall Officials: Işıl Özkoçak Turan, Prof., Study Director — Ministry of Health Ankara City Hospital
Locations (1):
- Ministry of Health Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No